CLINICAL TRIAL: NCT02434341
Title: Sleep Investigation in 3 Homogeneous Groups of Wake Mechanically Ventilated Patients in ICU: 1st Group - Septical Patients; 2nd Group - COPD Patients; 3rd Group - Surgical Patients, in Order to Define Common Sleep Features Within the Groups
Brief Title: Sleep in Critically Ill Patients on Mechanical Ventilation in ICU
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Yuliya Boyko, Yuliya Boyko, ph.d. student, MD, University of Southern Denmark
Other Study IDs: s-20140207G
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Polysomnographic Sleep Characteristics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- septic patients: wake septic patients on mechanical ventilation
- COPD patients: wake COPD patients on mechanical ventilation

SUMMARY:
15 patients with sepsis, 15 patients with COPD and 15 surgical patients will undergo polysomnographic sleep monitoring up to 24 hours in order to define if there are common sleep features within the groups

DETAILED DESCRIPTION:
It is an observational study in order to define if there are common polysomnographic sleep features within the following three groups of wake critically ill patients on mechanical ventilation in ICU: the group of septical patients, the group of patients with chronic obstructive pulmonary disease in exacerbation and the group of surgical patients without sepsis.

15 patients will be included in each group. They will undergo polysomnographic sleep monitoring during up to 24 hours.

Polysomnograms will be studies then in order to find out if there are common sleep characteristics within the homogeneous patient groups of critically ill.

ELIGIBILITY:
Inclusion Criteria:

* wake non-sedated patients
* mechanical ventilation

Exclusion Criteria:

* age < 18 years
* pregnant
* Glasgow Coma Scale < 11
* sedated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: wake
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
polysomnographic sleep features | polysomnographic sleep assessment during up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Boyko, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Intensive Care Unit, Odense University Hospital, Odense, Denmark